CLINICAL TRIAL: NCT04471922
Title: A Single-center, Randomized, Double-blinded, Placebo and Active Controlled Phase 1 Study to Evaluate the Safety and Pharmacology of Multiple Ascending Dose Administration of Anaprazole in Healthy Chinese Subjects
Brief Title: A Multiple Ascending High Dose Pharmacology Study of Anaprazole in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3571-CPK-1004
Record Dates: First submitted 2020-06-30; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anaprazole Sodium enteric-coated tablet (Experimental): "Multiple ascendinng dose, anaprazole 60mg QD(60mg QD group), 80mg QD(80mg QD group), 100mg QD(100mg QD group) , 7 days, fasting oral administration.
  "
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet
- Placebo (Placebo Comparator): Multiple dose, 1 tablet QD (60mg QD,80mg QD and 100mg QD group), 7 days, fasting oral administration.
  Interventions: Drug: Placebo
- Active controlled (rabeprazole) (Active Comparator): Multiple dose, rabeprazole 20mg QD (60mg QD,80mg QD and 100mg QD group), 7 days, fasting oral administration.
  Interventions: Drug: Active controlled (rabeprazole)

INTERVENTIONS:
Drug: Anaprazole Sodium enteric-coated tablet — Multiple ascendinng dose, anaprazole 60mg QD(60mg QD group), 80mg QD(80mg QD group), 100mg QD(100mg QD group) , 7 days, fasting oral administration.
  Arms: Anaprazole Sodium enteric-coated tablet
Drug: Placebo — Multiple dose, 1 tablet QD (60mg QD,80mg QD and 100mg QD group), 7 days, fasting oral administration.
  Arms: Placebo
Drug: Active controlled (rabeprazole) — Multiple dose, rabeprazole 20mg QD (60mg QD,80mg QD and 100mg QD group), 7 days, fasting oral administration.
  Arms: Active controlled (rabeprazole)

SUMMARY:
A single-center, randomized, double-blinded, placebo parallel controlled phase 1 study to evaluate the safety and pharmacokinetics/pharmacodynamics of multiple (7 days) ascending dose (60mg QD, 80mg QD, 100mg Qd) administrationof Anaprazole in healthy Chinese subjects. 45 subjects, 15 subjects for each dose group. In each dose group, 10 subjects take investigational drug (anaprazole), 2 subjects take active comparatory drug (rabeprazole), 3 subjects take placebo.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is capable of understanding and complying with protocol requirements, and signed and dated a written informed consent form voluntarily;
2. The subject is a Chinese health adult, aged 18 to 45 years, inclusive;
3. The subject weighed at least 50.0 kg and had a body mass index (BMI) between 19.0 kg/m^2 and 26.0 kg/m^2, inclusive;
4. Has clinical laboratory evaluations, vital signs and ECG testing (QTcF<450ms)within the reference range, and medical history and physicial examination results are normal. Participants with evaluations outside the reference range that are deemed not clinically significant by the investigator may be included at investigator discretion;
5. No medical history of allergy to proton pump inhibitors and no any other drug allergy history;
6. The subjects have a good lifestyle and can keep good communication with the investigators and comply with the requirements of clinical trial

Exclusion Criteria:

1. Has postural hypotension, gastrointestinal disease (gastric ulcer, gastritis and etc), liver disease, renal disease (nephritis, pyelonephritis and etc), and other disease or medical history of any other system (cardiovascular, respiratory, psychoneural, hematology, endocrinology and etc) ;
2. Has clinical significant abnormal electrolytes (especially hypopotassemia) in screening examination;
3. Has clinical significant ECG abnormal history or family history of long QT syndrome(Grandparents, parents and siblings);
4. Has rhinitis, allergic rhinitis, recurrent hemorrhinia, nasal deformity and abnormal nasal septum；
5. With positive result of drug screening test;
6. Female participants who are pregnant, breast-feeding or menstral period, or participants has no effective contraception method, or has pregnancy plan in 6 months;
7. Has received any drugs: acid-inhibitors, any priscription drug, herb medicine, non-prescription drugs and/or food suppliments (including vitamine) within 2 weeks before randomization;
8. Blood donation / blood loss ≥400 mL within 3 months, or participated any other clinical trials within 3 months;
9. Known Human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C antibody, and Treponema pallidum specific antibody test results were positive at screening;
10. Frequent alcoholics (drink more than 2 units of alcohol per day, 1 unit = 330 mL beer or 25 mL liquor or 125 mL wine), or took food or drinks with alcoholics 72 hours before randomization;
11. Has taken foods or drinks with xanthine(cafeine) or intensive excercise. Has taken foods or drinks that affect CYP3A4 (such as grapefruit or beverages containing grapefruit) within 14 days before administration of investigational drugs;
12. Smoke more than 5 pieces per week within 3 months before screening or can't stoping smok during study;
13. Any conditions in which considered by investigator not be appropriate to participate in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and serious adverse events as assessed by CTCAE v5.0 | From signing informed consent to study completion at 14 days after fist dose administration
  All adverse events will be monitored in each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China